CLINICAL TRIAL: NCT05739643
Title: A Phase 1/2 Clinical Study of Intravenous AAVrh10 Vector Expressing GALC in Krabbe Subjects Who Previously Received Hematopoietic Stem Cell Transplantation (REKLAIM)
Brief Title: Gene Transfer Clinical Trial for Infantile and Late Infantile Krabbe Disease Treated Previously With HSCT
Acronym: REKLAIM
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Forge Biologics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FBX-101-REKLAIM
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Krabbe Disease
Keywords: Leukodystrophy, Globoid Cell; Hereditary Central Nervous System Demyelinating Diseases; Brain Diseases, Metabolic, Inborn; Brain Diseases, Metabolic; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Sphingolipidoses; Lysosomal Storage Diseases, Nervous System; Leukoencephalopathies; Demyelinating Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Lipidoses; Lipid Metabolism, Inborn Errors; Lysosomal Storage Diseases; Metabolic Diseases; Lipid Metabolism Disorders
MeSH Terms: conditions — Leukodystrophy, Globoid Cell; Hereditary Central Nervous System Demyelinating Diseases; Brain Diseases, Metabolic, Inborn; Brain Diseases, Metabolic; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Sphingolipidoses; Lysosomal Storage Diseases, Nervous System; Leukoencephalopathies; Demyelinating Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Lipidoses; Lipid Metabolism, Inborn Errors; Lysosomal Storage Diseases; Metabolic Diseases; Lipid Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: Dose escalation study from a low dose to a high dose following safety review
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Low Dose FBX-101 (aka AAVrh.10-GALC) (Experimental): N=3 patients with Infantile or Late Infantile Krabbe disease will receive a single infusion at the low dose
  Interventions: Biological: FBX-101
- Cohort 2 - High Dose FBX-101 (aka AAVrh.10-GALC) (Experimental): N=3-6 patients with Infantile or Late Infantile Krabbe disease will receive a single infusion at the high dose
  Interventions: Biological: FBX-101

INTERVENTIONS:
Biological: FBX-101 — A replication-deficient adeno-associated virus gene transfer vector expressing the human galactocerebrosidase (GALC) cDNA will be delivered one-time through a venous catheter inserted into a peripheral limb vein.
  Other Names: AAVrh.10-hGALC

SUMMARY:
This is a non-blinded, non-randomized dose escalation study of intravenous FBX-101 in which subjects will receive a single infusion of an adeno-associated virus gene therapy product, after more than 21 days of the HSCT (UCBT preferred HSCT source). Data from previously transplanted patients with infantile and late infantile Krabbe disease will be used as a comparator group.

DETAILED DESCRIPTION:
The FBX-101-REKLAIM study has been modified on Q4 2023 to allow a broader patient recruitment of infantile and late infantile Krabbe patients. The updated REKLAIM study merges the recruitment populations of the previous FBX-101-RESKUE clinical trial (NCT04693598) and the FBX-101-REKLAIM clinical trial (NCT05739643).

ELIGIBILITY:
Inclusion Criteria:

1. Group Infantile Krabbe: Subjects who are going to be transplanted or have already been transplanted for asymptomatic infantile onset Krabbe disease with initial diagnosis based on:

   1. Galactocerebrosidase (GALC) activity levels in leukocytes compatible with the diagnosis of infantile Krabbe disease; AND AT LEAST ONE OF THE FOLLOWING:
   2. Psychosine levels predictive of infantile onset by Dried Blood Spot (DBS); OR
   3. Imaging or neurophysiological findings consistent with Krabbe disease (CSF, MRI, NCV, ABR); OR
   4. Two GALC mutations predictive to result in infantile onset phenotype.
2. Group Late Infantile Krabbe: Subjects who are going to be transplanted or have already been transplanted for symptomatic late infantile onset Krabbe with initial diagnosis based on:

   1. Galactocerebrosidase (GALC) activity levels in leukocytes compatible with the diagnosis of late infantile Krabbe disease; AND AT LEAST ONE OF THE FOLLOWING:
   2. Psychosine levels predictive of late infantile onset by DBS; OR
   3. Imaging or neurophysiological findings consistent with Krabbe disease (CSF, MRI, NCV, ABR); OR
   4. Two GALC mutations predictive to result in late infantile onset phenotype; OR
   5. Neurological/developmental exam findings consistent with late infantile Krabbe disease
3. Participants must be considered candidates for HSCT or have received HSCT at least 21 days prior to dosing date
4. For patients already transplanted and followed for more than 3 months chimerism should reflect at least 30% of myeloid cells from the donor by month 3 post-transplant, from 30 to 10% between 3 months and one year post-transplant or 10% by one year post-transplant.
5. Participant must have adequate organ function at time of screening or evaluation as measured by:

   1. Ejection fraction of > 50% by echocardiogram or other appropriate study without evidence of pulmonary hypertension.
   2. Pulmonary evaluation testing demonstrating resting pulse oximeter > 95% on room air.
6. Absence of active aspiration
7. Participant's parents or legal guardian consent to participate in the study and provide informed consent according to IRB/IEC guidelines prior to any study procedures being performed
8. Parent(s) and/or legal guardian able to comply with the clinical protocol

Exclusion Criteria:

1. Immunoassay with total anti-AAV10 antibody titers of >1:100. This criterion will not apply to children screened before they have received HSCT or for children who sign the inform consent within 6 months from HSCT. In children who test positive to anti-AAV10 antibody with titers of >1:100 under this exception, the ISR regime proposed by the PI and approved/modified by the ISR committee may include immunosuppressive drugs that prevent the potential development of a secondary immune response to AAVrh10 after FBX-101 administration.
2. History of prior treatment with a gene therapy product
3. Motor function evaluated by age with PDMS-II by a study physical therapist:

   a. Inability to hold head for patients older than 5 months; b. Inability to sit independently for patients older than 12 months; c. Inability to walk with assistance for patients older than 24 months.
4. In patients that sign the informed consent before HSCT or up to 90 days post-HSCT, abnormalities in white count, hemoglobin and platelets found from conditioning regime to Day -1 (the day before FBX-101 administration) will be evaluated by the PI (with referral to the DSMB if indicated). If abnormal, they will not be considered an exclusion criteria if the PI considers they are consistent with expected consequences of the HSCT (and related management) and upon confirmation they were not present before commencement of the conditioning regime.
5. Grade 2 or higher abnormalities in LFTs, bilirubin, creatinine, white count, hemoglobin, platelets, PT/INR and PTT according to latest version of CTCAE
6. Presence of any neurocognitive deficit, motor deficit, or brain damage not attributable to Krabbe disease
7. Signs of active infections or disease from cytomegalovirus, adenovirus, EBV, hepatitis B or C, and HIV or other viruses excluding rhinovirus from RVP and asymptomatic norovirus presence in stool. Patients showing HIV positive results will be excluded from the study.
8. Active bacterial or fungal infection documented the preceding 7 days.
9. Presence of any contraindication for MRI or lumbar puncture (LP)
10. Use of any investigational product prior to study enrollment or current enrollment in another study that involves clinical interventions
11. Immunizations with live viruses in the 30 days prior to immune suppression
12. Active acute Graft Versus Host Disease (GvHD) Grade II or higher according to modified Glucksberg criteria (Przepiorka et al., 1995) or active, moderate or severe, chronic GvHD according to revised NIH criteria (Jagasia et al., 2015)
13. Any other medical condition, serious intercurrent illness, other genetic condition or extenuating circumstance that, in the opinion of the PI, would preclude participation in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by incidence and severity of adverse events and serious adverse events that are attributed to FBX-101 | 24 months

SECONDARY OUTCOMES:
Efficacy as assessed by improvement of gross motor function as measured longitudinally by PDMS-2, BOT-3, or by GMFM-88, depending on the age, compared to patients receiving HSCT only | 12 months and 24 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's Hospital of Orange County (CHOC), Orange, California
  - University of Michigan Hospitals - Michigan Medicine, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bascou N, DeRenzo A, Poe MD, Escolar ML. A prospective natural history study of Krabbe disease in a patient cohort with onset between 6 months and 3 years of life. Orphanet J Rare Dis. 2018 Aug 9;13(1):126. doi: 10.1186/s13023-018-0872-9. PMID 30089515
- [Background] Beltran-Quintero ML, Bascou NA, Poe MD, Wenger DA, Saavedra-Matiz CA, Nichols MJ, Escolar ML. Early progression of Krabbe disease in patients with symptom onset between 0 and 5 months. Orphanet J Rare Dis. 2019 Feb 18;14(1):46. doi: 10.1186/s13023-019-1018-4. PMID 30777126
- [Background] Escolar ML, Poe MD, Provenzale JM, Richards KC, Allison J, Wood S, Wenger DA, Pietryga D, Wall D, Champagne M, Morse R, Krivit W, Kurtzberg J. Transplantation of umbilical-cord blood in babies with infantile Krabbe's disease. N Engl J Med. 2005 May 19;352(20):2069-81. doi: 10.1056/NEJMoa042604. PMID 15901860
- [Background] Escolar ML, West T, Dallavecchia A, Poe MD, LaPoint K. Clinical management of Krabbe disease. J Neurosci Res. 2016 Nov;94(11):1118-25. doi: 10.1002/jnr.23891. PMID 27638597
- [Background] Rafi MA, Luzi P, Wenger DA. Conditions for combining gene therapy with bone marrow transplantation in murine Krabbe disease. Bioimpacts. 2020;10(2):105-115. doi: 10.34172/bi.2020.13. Epub 2020 Mar 24. PMID 32363154
- [Background] Yoon IC, Bascou NA, Poe MD, Szabolcs P, Escolar ML. Long-term neurodevelopmental outcomes of hematopoietic stem cell transplantation for late-infantile Krabbe disease. Blood. 2021 Apr 1;137(13):1719-1730. doi: 10.1182/blood.2020005477. PMID 33150395
- [Background] Wright MD, Poe MD, DeRenzo A, Haldal S, Escolar ML. Developmental outcomes of cord blood transplantation for Krabbe disease: A 15-year study. Neurology. 2017 Sep 26;89(13):1365-1372. doi: 10.1212/WNL.0000000000004418. Epub 2017 Aug 30. PMID 28855403
- [Background] Gupta A, Poe MD, Styner MA, Panigrahy A, Escolar ML. Regional differences in fiber tractography predict neurodevelopmental outcomes in neonates with infantile Krabbe disease. Neuroimage Clin. 2014 Sep 26;7:792-8. doi: 10.1016/j.nicl.2014.09.014. eCollection 2015. PMID 25844309
- [Background] Escolar ML, Poe MD, Smith JK, Gilmore JH, Kurtzberg J, Lin W, Styner M. Diffusion tensor imaging detects abnormalities in the corticospinal tracts of neonates with infantile Krabbe disease. AJNR Am J Neuroradiol. 2009 May;30(5):1017-21. doi: 10.3174/ajnr.A1476. Epub 2009 Apr 22. PMID 19386732
- [Background] Bradbury AM, Bagel J, Swain G, Miyadera K, Pesayco JP, Assenmacher CA, Brisson B, Hendricks I, Wang XH, Herbst Z, Pyne N, Odonnell P, Shelton GD, Gelb M, Hackett N, Szabolcs P, Vite CH, Escolar M. Combination HSCT and intravenous AAV-mediated gene therapy in a canine model proves pivotal for translation of Krabbe disease therapy. Mol Ther. 2024 Jan 3;32(1):44-58. doi: 10.1016/j.ymthe.2023.11.014. Epub 2023 Nov 11. PMID 37952085
- [Result] Greco MR, Lopez MA, Beltran-Quintero ML, Tuc Bengur E, Poe MD, Escolar ML. Infantile Krabbe disease (0-12 months), progression, and recommended endpoints for clinical trials. Ann Clin Transl Neurol. 2024 Dec;11(12):3064-3080. doi: 10.1002/acn3.52114. Epub 2024 Nov 5. PMID 39499628